CLINICAL TRIAL: NCT04442061
Title: Autism Spectrum Disorders: Double Blind Randomized Placebo-control Active Pilot Study of Transcranial Magnetic Stimulation Applied to the Superior Temporal Sulcus
Acronym: STIMAUT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation de France (Other); Fondation Malakoff Médéric (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APHP191009
Record Dates: First submitted 2020-04-20; First posted 2020-06-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Autism Spectrum Disorders
Keywords: transcranial magnetic stimulation; superior temporal sulcus
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Transcranial Magnetic Stimulation; Neuronavigation; Eye-Tracking Technology

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active transcranial magnetic stimulation (Active Comparator): excitatory TMS will be applied to the right posterior STS
  Interventions: Device: Transcranial magnetic stimulation; Device: MRI; Device: Neuronavigation; Device: Eye-tracking; Genetic: Salivary samples; Other: Clinical scales
- Sham transcranial magnetic stimulation (Sham Comparator): The sham TMS follows the same procedure of the active TMS without stimulating cortical tissue
  Interventions: Device: Transcranial magnetic stimulation; Device: MRI; Device: Neuronavigation; Device: Eye-tracking; Genetic: Salivary samples; Other: Clinical scales

INTERVENTIONS:
Device: Transcranial magnetic stimulation — Before the stimulation, identification of a motor "hotspot" and active motor threshold (AMT) will be performed. The TMS will be applied on the intermittent theta-burst modality (iTBS), i. e., 2 s of TBS trains (30 pulses) repeated every 10 s for 190 s, with a total number of 600 pulses (Huang et al, 2005). The whole TMS session, including preparation, will last up to 1h.
  The sham TMS follows the same procedure of the active TMS without stimulating cortical tissue
Device: MRI — Anatomical and functional images will be acquired and review by an experienced neuro-radiologist.
Device: Neuronavigation — The neuronavigation system will allow to guide the stimulation using the individual anatomical MRI acquired with MRI, and to record the position and orientation of the coil during successive stimulations
Device: Eye-tracking — Eye movements and follow a person's gaze will be recorded during visualization of stimuli presented in the screen by analyzing images of the eye captured by an infrared camera
Genetic: Salivary samples — The DNA will be extracted from the salivary sample to genotyping analyses on the BDNF (Val66Met) and COMT (Val158Met) polymorphism
Other: Clinical scales — CGI, E-CAR and ABC will be used for behavior and clinical evaluation

SUMMARY:
Difficulties in social interactions are the core feature of autism spectrum disorder (ASD) and are characterized by abnormal social perception, mainly concerning eye gaze. Anatomo-functional abnormalities within the superior temporal sulcus (STS), a key region of the social brain, have been described in ASD. The investigators had recently shown that it is possible to modulate the neural activity of the STS with transcranial magnetic stimulation (TMS) with an impact on social perception, measured by eye-tracking. In the context of ASD, stimulation of the STS with excitatory TMS could lead to an improvement in social perception, which would open up new therapeutic strategies. The purpose of this double-blind, randomized, placebo-controlled study is to apply a therapeutic TMS protocol (10 daily sessions) at the right STS in young adults with ASD to improve their social behavior, objectively measured using eye-tracking.

DETAILED DESCRIPTION:
Autism Spectrum Disorders (ASD) are neuro-developmental disorders presumably related to neural circuit alterations. The symptoms, that start very early in development and persist through adulthood, can lead to severe handicap. Even though a wide variety of clinical severity exists, difficulties in social interactions are a core feature of ASD. These difficulties are characterized by social perception abnormalities, manifested mainly through abnormal eye contact. Such abnormalities have been largely confirmed in the last decade by eye-tracking studies, which allow objective and quantitative investigation of gaze behaviour. Studies with adults and children with ASD during visualization of social scene have shown a lack of preference for socially relevant information, mainly faces and eyes.

In the typically developing brain, socially relevant information is processed within a specific network, called the social brain. Functional MRI (fMRI) activation studies have shown the implication of a key region of the social brain, namely the superior temporal sulcus (STS), is in processing social information, ranging from the perception of eyes, faces and voices to the more complex processes of social cognition. Over the last decades, brain imaging studies investigating the neuro basis of ASD have consistently described anatomical and functional abnormalities within the social brain, particularly within the STS Currently there are important limitations in the therapeutic interventions available for ASD. Pharmacological treatments are only indicated for psychiatric comorbidity and has no impact on ASD core manifestations. Behavioural interventions, on the other hand, are generally expensive, time-consuming and have modest results. In more recent years non-invasive neuromodulation techniques, such as Transcranial Magnetic Stimulation (TMS), have raised hope as effective tool to address ASD core manifestations. Indeed, modulating the neural activity of STS with an impact on social perception opens new therapeutic perspectives in ASD. The effect of TMS on social behaviour has been recently showed by a study from our lab. Following an inhibition of the right STS by inhibitory TMS, healthy volunteers look less at the eyes of the characters during the visualization of social scenes.

In this context, the main objective of this study is to investigate the effect of repetitive session of TMS applied to the STS on social perception in patients with ASD. In addition, the investigators aim to research the impact of putative changes in social perception in broader social behaviour using clinical scales. Finally, the investigators aim to research putative changes in brain functioning at rest by measuring rest cerebral blood flow using Arterial Spin Labeling (ASL)-MRI before and after TMS. This is a double-blind, randomized, placebo-controlled therapeutic trial, ultimately aiming to improve broader social behaviour.

For that purpose, the investigators will include in the present study 20 participants with non-syndromic ASD aged from 18 to 25 years old. Social perception will be measured using an eye-tracking during passive visualization of social stimuli. All patients will undergo an MRI for neuronavigation purposes and to obtain rest cerebral blood flow measures using arterial spin labelling MRI sequence, as well as clinical scales to evaluate their global social behavior: clinical global impressions (CGI), "évaluation des comportements autistiques revise" (ECA-R) and autism behavior checklist (ABC). The 20 patients will be automatically randomized in the active TMS arm (n = 10), or in the placebo arm (n = 10). Patients will undergo 10 sessions of TMS applied to the posterior part of the right superior STS, from Monday to Friday for two consecutive weeks. Following the 10 sessions, evaluations will be performed: 5 days, 1 month and 3 months after the end of the treatment.

The investigators expect that stimulation of the posterior part of the STS, a region shown to be strongly implicated in processing social information, mainly from the eyes, would lead to an increase in eye-gaze perception and thus promote access to social cues necessary for adapted broader social behavior. If so, TMS could be further considered as an alternative therapeutical intervention in ASD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient diagnosed with ASD according to DSM-V and ADI-R
* Patient aged 17 to 25
* Patient apt to undergo an MRI
* Patient affiliated with a social security system or beneficiary of such system
* Informed consent signed by the patient or his legal guardian.

Exclusion Criteria :

* Presence of a somatic pathology
* Presence of a neurological pathology
* Presence of epilepsy, history of seizure.
* Initiation, discontinuation or modification of neuroleptics or benzodiazepines treatment in the previous month
* Contraindication to MRI (pacemaker, intracorporeal metallic foreign body, metal worker)
* Contraindication to the use of TMS (epilepsy and family epilepsy, presence of craniotomy scar, pacemaker or pacemaker, intraocular or intracerebral metallic foreign body, cochlear implant, cardiac valve or metallic surgical arterial material, metallic material capable of concentrating radio frequency pulses)
* Pregnancy and breast-feeding
* Participation in another pilot study or clinical trial that does not allow participation in this protocol.

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes gaze pattern to the eyes | Until 3 months after iTBS sessions
  Changes number of fixations to the eyes measured by eye-tracking during passive visualization of social scenes following the 10 iTBS sessions applied to the right pSTS compared to baseline measures.

SECONDARY OUTCOMES:
Autistic Behavior Checklist (ABC) scale at v1 | 5 days before iTBS sessions
  Evaluate social behavior and autistic symptoms (Lower score = 0 Higher score mean worse outcome = 174)
Autistic Behavior Checklist (ABC) scale at v2 | 5 days after iTBS sessions
  Evaluate social behavior and autistic symptoms (Lower score = 0 Higher score mean worse outcome = 174)
Autistic Behavior Checklist (ABC) scale at v3 | 1 month after iTBS sessions
  Evaluate social behavior and autistic symptoms (Lower score = 0 Higher score mean worse outcome = 174)
Autistic Behavior Checklist (ABC) scale at v4 | 3 months after iTBS sessions
  Evaluate social behavior and autistic symptoms (Lower score = 0 Higher score mean worse outcome = 174)
"Evaluation des comportements Autistiques révisée" (ECA-R) scale at v1 | 5 days before iTBS sessions
  Evaluate social behavior and autistic symptoms (Lower score = 0 Higher score mean worse outcome = 116)
"Evaluation des comportements Autistiques révisée"(ECA-R) scale at v2 | 5 days after iTBS sessions
  Evaluate social behavior and autistic symptoms (Lower score = 0 Higher score mean worse outcome = 116)
"Evaluation des comportements Autistiques révisée" (ECA-R) scale at v3 | 1 month after iTBS sessions
  Evaluate social behavior and autistic symptoms (Lower score = 0 Higher score mean worse outcome = 116)
"Evaluation des comportements Autistiques révisée" (ECA-R) scale at v4 | 3 months after iTBS sessions
  Evaluate social behavior and autistic symptoms (Lower score = 0 Higher score mean worse outcome = 116)
Clinical Global Impression (CGI) scale at v1 | 5 days before iTBS sessions
  global functioning (Lower score = 1 Higher score mean worse outcome=16)
Clinical Global Impression (CGI) scale at v2 | 5 days after iTBS sessions
  global functioning (Lower score = 1 Higher score mean worse outcome=16)
Clinical Global Impression (CGI) scale at v3 | 1 month after iTBS sessions
  global functioning (Lower score = 1 Higher score mean worse outcome=16)
Clinical Global Impression (CGI) scale at v4 | 3 months after iTBS sessions
  global functioning (Lower score = 1 Higher score mean worse outcome=16)
Changes in rest brain fonctionning at v1 | 5 days before iTBS sessions
  by measuring whole brain cerebral blood flow at rest using MRI-ASL
Changes in rest brain fonctioning at v2 | 5 days after iTBS sessions
  by measuring whole brain cerebral blood flow at rest using MRI-ASL
Changes in rest brain fonctioning at v4 | 3 months after iTBS sessions
  by measuring whole brain cerebral blood flow at rest using MRI-ASL
Putative changes on brain functional connectivity at rest at V1 | 5 days before iTBS sessions
  by using the resting state sequence using MRI-ASL
Putative changes on brain functional connectivity at rest at V2 | 5 days after iTBS sessions
  by using the resting state sequence using MRI-ASL
Putative changes on brain functional connectivity at V4 | 3 months after iTBS sessions
  by using the resting state sequence using MRI-ASL
Anatomical connectivity abnormalities | At V1 : 5 days before iTBS sessions
  by using the diffusion tensor imaging sequence (DTI) using MRI-ASL
BDNF/COMT polymorphisms | 5 days after baseline
  Research of BDNF/COMT polymorphisms on salivary samples

CONTACTS AND LOCATIONS:
Overall Officials: Monica ZILBOVICIUS, Study Chair — INSERM ERL "Trajectoires Developpementales en Psychiatrie"
Locations (1):
- Hôpital Necker Enfants Malades - Service de radiologie pédiatrique, Paris, France

IPD SHARING:
Plan to Share IPD: No